CLINICAL TRIAL: NCT03460938
Title: The Effect of Remote Ischemic Preconditioning on Postoperative Myocardial Ischemia in Pancreatic Surgery: a Randomized Controlled Trial
Brief Title: Remote Ischemic Preconditioning and Postoperative Myocardial Ischemia
Acronym: MICOLON2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, Principal Investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL57818.100.16
Record Dates: First submitted 2017-03-29; First posted 2018-03-09 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Myocardial Ischemia; Inflammatory Response
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC (Experimental)
  Interventions: Procedure: Remote ischemic preconditioning
- Control (No Intervention)

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — RIPC: 3 periods of 5 minutes of ischemia followed by 5 minutes of reperfusion are created by inflating a blood pressure cuff on the upper extremity after induction of anesthesia and prior to surgery.
  Arms: RIPC

SUMMARY:
High-risk abdominal surgery is frequently complicated by postoperative complications, such as sepsis, pneumonia or anastomotic dehiscence. Asymptomatic myocardial injury after abdominal surgery (MINS) predicts non-cardiac complications. The etiology of MINS in abdominal surgery patients is unknown. Remote ischemic preconditioning (RIPC) is a physiologic mechanism that exposes tissues to brief periods of non-lethal ischemia and reperfusion, creating resistence for future serious ischemic insults. RIPC in patients after cardiac or aortic surgery is associated with a protective effect on the heart. The effect of RIPC in abdominal surgery patients is unknown.

Objective of the study: To determine the effect of RIPC on MINS in patients after pancreatic sugery.

Study design: Randomised controlled parallel group mono-center pilot study.

Study population: 90 adult patients scheduled for elective pancreaticoduodenectomy in St. Antonius Hospital (45 in the intervention group and 45 in the control group).

Intervention: RIPC: 3 periods of 5 minutes of ischemia followed by 5 minutes of reperfusion are created by inflating a blood pressure cuff on the upper extremity after induction of anesthesia and prior to surgery. In the control group a non-inflated blood pressure cuff is placed on the upper extremity for 30 minutes.

Primary study parameters/outcome of the study: Maximum postoperative concentration of high-sensitive cardiac troponin T.

Secondary study parameters/outcome of the study: Markers of inflammatory, intestinal and renal injury, postoperative complications during 30 days, length of stay and hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Elective pancreaticoduodenectomy
* Age >18

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative myocardial injury. | 48 hours
  Maximum postoperative concentration of high-sensitive cardiac troponin T.

SECONDARY OUTCOMES:
Inflammatory response | 48 hours
  Markers of inflammation (IL6)
Postoperative complications | 30 days
  Postoperative cardiac and noncardiac complications

CONTACTS AND LOCATIONS:
Overall Officials: Peter Noordzij, MD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reniers T, Rettig T, van Zeggeren L, Dijkstra I, Prinsze K, Molenaar I, van Santvoort H, Cremer O, Vernooij L, Noordzij P. Is chronic inflammation a risk factor for perioperative myocardial injury or heart failure in pancreatic surgery patients? BJA Open. 2025 May 19;14:100417. doi: 10.1016/j.bjao.2025.100417. eCollection 2025 Jun. PMID 40491666
- [Derived] van Zeggeren L, Visser RA, Vernooij LM, Dijkstra IM, Bosma M, Molenaar Q, van Santvoort HC, Noordzij PG. The effect of remote ischaemic preconditioning on postoperative cardiac and inflammatory biomarkers in pancreatic surgery: a randomized controlled trial. BJS Open. 2021 Mar 5;5(2):zrab015. doi: 10.1093/bjsopen/zrab015. PMID 33893738